CLINICAL TRIAL: NCT07213141
Title: Incidence of Graves' Disease After COVID-19 Vaccination: a Retrospective Analysis
Brief Title: Incidence of Graves' Disease After COVID-19 Vaccination
Status: Active, not recruiting | Type: Observational
Sponsor: Laura ICONARU (Other)
Responsible Party: Sponsor-Investigator, Laura ICONARU, Head of Endocrinology department, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Graves
Record Dates: First submitted 2025-05-19; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Graves Disease
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 'de novo' Graves' disease: All patients who developed 'de novo' Graves' disease between March 2020 (the beginning of the COVID-19 epidemic in Belgium) and October 2022
  Interventions: Other: Data extraction

INTERVENTIONS:
Other: Data extraction — Data extraction from medical records

SUMMARY:
It is well known that an infection can be a triggering factor for the development of autoimmune thyroid disease. The COVID-19 pandemic was an example of this, with several reports of both subacute thyroiditis as well as Graves' disease occurring after experiencing SARS-CoV-2 disease. There have also been cases of Graves' disease reported after COVID-19 vaccination administration (<4 weeks between the vaccine and the development of hyperthyroidism). However, the current evidence is of low quality and consists mainly of case reports. A search strategy on October 3, 2022, in the medical database PubMed could only retain one retrospective study on this subject. In this study by di Filippo et al., approximately 64 new cases of Graves' disease with hyperthyroidism were identified in the Milan region, Italy, in the year 2021, of which 20 patients had an onset within 4 weeks following COVID vaccine administration (31.2%).

The investigators would like to increase the knowledge about the possible link between COVID-19 (both the disease and the vaccination) and Graves' disease, by means of a case-control analysis of all 'de novo' cases of Graves' hyperthyroidism described in the C.H.U. Brugmann. The investigators want to investigate whether Graves' disease after vaccination would be clinically different from the "classic" Graves' disease, thereby describing factors such as the duration of the disease, the level of thyroid-stimulating immunoglobulins (TSI), the percentage of T3-dominant Graves' disease, or the dose of thyreostatics (such as strumazole) required to control the disease.

ELIGIBILITY:
Inclusion Criteria:

All patients who developed 'de novo' Graves' disease between March 2020 (the beginning of the COVID-19 epidemic in Belgium) and October 2022.

Exclusion Criteria:

* Pregnancy
* Pre-existing Graves' disease (before March 2020)
* Diagnosis of other thyroid disease, such as subacute or painless destructive thyroiditis
* Use of thyroid-interfering drugs, such as lithium, amiodarone or immune checkpoint inhibitor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who developed 'de novo' Graves' disease between March 2020 (the beginning of the COVID-19 epidemic in Belgium) and October 2022. These patient cases will be identified based on the biochemical-radiological factors diagnostic for "classic" Graves' disease, i.e., hyperthyroidism in the context of positivity for TSI and/or homogeneous captation on thyroid scintigraphy
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographic data | 2 years
  Age, gender and smoking
COVID-19 infection (yes/no) | 2 years
  Evidence for COVID-19 infection, based on emergency room consultation, hospitalization for COVID-19, positive PCR testing or CT scan
COVID-19 vaccination status | 2 years
  Timing, type and dosing of COVID-19 vaccine administration
TSH levels | 2 years
  Blood levels of thyroid-stimulating hormone (Thyroid hormone)
Free thyroxine levels | 2 years
  Free thyroxine blood levels (Thyroid hormone)
Free T3 levels | 2 years
  Free T3 blood levels (Thyroid hormone)
TSI levels | 2 years
  Blood levels of thyroid-stimulating immunoglobulin (thyroid autoantibodies)
Anti-thyroperoxidase levels | 2 years
  Thyroid autoantibodies levels (thyroid autoantibodies)
Anti-thyroglobulin levels | 2 years
  Thyroid autoantibodies levels (thyroid autoantibodies)
Conclusions of the Thyroid ultrasound examination | 2 years
Conclusions of the Thyroid scintigraphy examination | 2 years
Anti-thyroid treatment | 2 years
  Narrative description of anti-thyroid treatments, if any

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen de Filette, MD, Study Director — CHU Brugmann
Locations (3):
- Belgium (3):
  - CHU St Pierre, Brussels
  - CHU Brugmann, Brussels
  - UZ Brussel, Jette

IPD SHARING:
Plan to Share IPD: No